CLINICAL TRIAL: NCT04462081
Title: Non Alcoholic Fatty Liver Disease and Coronary Heart Disease in Type 2 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rohit Loomba, Associate Professor of Clinical Medicine, University of California, San Diego
Other Study IDs: NAFLD and CHD in Diabetes
Record Dates: First submitted 2014-12-17; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2016-09

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — There is a separate optional component of the study where subjects will be asked to donate a blood sample for genetic research.Subjects will be offered the opportunity to review, discuss and sign the consent at their scheduled visit. All questions will be answered at this time and throughout the study. Declining to give a genetic sample does not prohibit the participant from participating in the study. The biospecimen collected as part of this study will be kept in Dr. Loomba's locked research freezer at the Clinical Teaching Facility (CTF-building A).These samples and data may be stored for 50 years to be used at a later date for investigation of new novel biomarkers. This will be made clear to the patient during the consent process.
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the feasibility in diabetics in a primary care setting of screening for NAFLD and advanced fibrosis, by using non-invasive magnetic resonance imaging (MRI) to estimate the hepatic proton density fat fraction (MRI-PDFF) and magnetic resonance elastography (MRE) to estimate hepatic stiffness.

DETAILED DESCRIPTION:
This is a prospective cohort study consisting of a one-time visit by diabetic patients with optional following liver biopsy. The aim of the study is to evaluate whether liver fat fraction and liver stiffness, as determined by magnetic resonance imaging, are associated with subclinical cardiovascular disease, as evaluated by coronary artery calcium scan in diabetics. During the visit, patients will undergo review of medical history, vitals (including body mass index, blood pressure), physical exam, blood work, urine collection, ECG, magnetic resonance imaging (MRI), including MR proton density fat fraction (MRI-PDFF) and MR elastography, ultrasound using acoustic radiation force impulse (ARFI) imaging, and computed tomography (CT) scan for coronary artery calcium scoring. Blood work will be sent for labs relevant to traits of metabolic syndrome including markers for diabetes (hemoglobin A1C, fasting glucose) and hyperlipidemia (lipid panel). Serum, plasma and whole blood will be stored for future studies. Results from history, physical exam, and radiographic imaging will be analyzed and if they indicate the presence of nonalcoholic steatohepatitis, patients will be offered an optional liver biopsy for further assessment. All patients will be invited to continue in the study and have follow-up visits every two years for a total duration of the study of 5 years.

ELIGIBILITY:
Inclusion criteria:

* Adults, age 21 or above, with diagnosis of T2DM according to the American Diabetes Association (ADA) clinical practice recommendations.
* T2DM is defined according to American Diabetes Association (ADA) clinical practice recommendations if one of the following criteria is met:

  * Diabetes symptoms (polyuria, polydipsia, polyphagia, increased fatigue, weight loss, blurred vision) exist and casual plasma glucose ≥200 mg/dl (11.1 mmol/l) OR
  * Fasting plasma glucose (FPG) ≥126 mg/dl (7.0 mmol/l); OR
  * Plasma glucose ≥200 mg/dl (11.1 mmol/l) during a 75-g oral glucose tolerance test (OGTT) (25).
* If any of these test results occur, testing should be repeated on a different day to confirm the diagnosis. OR

  * hemoglobin A1C (HbA1C) ≥6.5% (26).
* The subject is fully informed and willing and able to perform all the procedures specified in the protocol and signed a written informed consent to participate

Exclusion criteria:

* Documented history of cardiovascular disease (CVD), such as acute coronary syndrome (ST elevation myocardial infarction, non-ST elevation myocardial infarction, unstable angina), stable angina, history of angioplasty or stent placement, cerebrovascular disease (ischemic or hemorrhagic stroke), and peripheral vascular disease.
* History of congestive heart failure
* Evidence of other causes of chronic liver disease

  * Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg).
  * Previous or current infection with Hepatitis C as defined by presence of hepatitis C virus Ab in serum (anti-HCV Ab).
  * Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
  * Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.
  * Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.
  * Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
  * Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D.
  * Drug-induced liver disease as defined on the basis of typical exposure and history.
  * Bile duct obstruction as shown by imaging studies.
* History of gastrointestinal bypass surgery or ingestion of medications known to produce steatosis, such as corticosteroids, high-dose estrogen, tamoxifen, methotrexate, amiodarone or tetracycline in the previous 6 months.
* Evidence of cirrhosis or previously known cirrhosis based on the results from previous liver biopsy or history of portal hypertension presented by ascites, hepatic encephalopathy or varices
* Absence of regular and/or excessive use of alcohol(defined as >30g/day for males and >15g/day for females) for a period longer than 2 years at any times in the last 10 years
* Serum creatinine> 1.5 mg/dL
* The subject is a pregnant or nursing female
* Contraindications to computed tomography (CT) or magnetic resonance imaging (MRI):

  * The subject has any contraindication to MR imaging, such as patients with cardiac pacemaker or defibrillator, neurostimulator, intravascular stents, coils, valves, surgical clips, implanted electronic infusion pump, ferromagnetic foreign body or other conditions that would preclude proximity to a strong magnetic field.
  * The subject has a history of extreme claustrophobia.
  * The subject cannot fit inside the MRI or CT machine

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, age 21 or above, with diagnosis of T2DM according to the American Diabetes Association (ADA) clinical practice recommendations.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Liver Fat as Measured by MRI-PDFF | Baseline
  Evaluation of liver fat fraction and liver stiffness, as determined by magnetic resonance imaging, are associated with subclinical cardiovascular disease, as evaluated by coronary artery calcium scan in diabetics

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No